CLINICAL TRIAL: NCT03798886
Title: Comparison of Clinical Results of Frozen Embryo Transfer in Natural and Modified Natural Cycles
Brief Title: Success Rate Natural Cycles Versus Modified Natural Cycles in Frozen Embryos
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: ATADEK-2018/20
Record Dates: First submitted 2019-01-07; First posted 2019-01-10 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Infertility, Female
Keywords: Frozen embryo replacement, IVF success, ovarian stimulation
MeSH Terms: conditions — Infertility, Female | interventions — Embryo Transfer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patient blood sample for hormonal assay
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Natural frozen embryo transfer group: In this group all embryos will be frozen when transfer planned sonographic follicle diameter measured. After spontaneous ovulation, embryo transfer will be planned. Luteal phase support will not be used.
  Interventions: Other: natural cycle; Other: modified natural cycle; Other: embryo transfer
- modified natural embryo transfer group: In this group all embryos will be frozen when transfer planned sonographic follicle diameter measured. When follicle diameter is 16-17 mm we will apply hCG (recombinant hCG). After ovulation, embryo transfer will be done. Luteal phase support will not be used.
  Interventions: Other: natural cycle; Other: modified natural cycle; Other: embryo transfer

INTERVENTIONS:
Other: natural cycle — When follicle is ready for ovulation, we will use this injection by intra-dermal route
  Other Names: natural LH surge
Other: modified natural cycle — we will use that drug in the natural modified transfer group after embryo transfer
  Other Names: recombinant hcg
Other: embryo transfer — we will do transfer when the endometrium is ready
  Other Names: frozen embryo transfer

SUMMARY:
There has been a recent significant increase in the frozen embryo replacement (FER) cycles due to freeze-all cycles to decrease the risk of ovarian hyperstimulation syndrome. Now a days making frozen embryo transfers (FETs) a viable alternative to fresh embryo transfer

DETAILED DESCRIPTION:
There has been a recent significant increase in the frozen embryo replacement (FER) cycles due to freeze-all cycles to decrease the risk of ovarian hyperstimulation syndrome. Now a days making frozen embryo transfers (FETs) a viable alternative to fresh embryo transfer, with reports from observational studies and randomized controlled trials suggesting that:

1. The endometrium in stimulated cycles is not optimal for implantation
2. Pregnancy rates are increased following FET
3. Perinatal outcomes are less affected after FET
4. Preimplantation genetic screening We will follow only natural and modified natural cycles patients. Spontaneous ovulation will documented with hormonal and sonographic monitoring. Hormonal monitoring are including estradiol and luteinizing hormone (LH). Sonographic monitoring is including follicule diameter (16-20 mm). At modified natural cycles we will use hCG triggering for ovulation approximately 16-20 mm diameter.

We will compare success rate between natural and modified natural cycles

ELIGIBILITY:
Inclusion Criteria:

* Patient who are admitted to the IVF center and who will be transferred to frozen embryos.
* Infertile women under 40 years of age who accepted this study.
* Unexplained infertilite couple.
* All ovulatory patient.
* Male factor.
* Tubal factor.

Exclusion Criteria:

* Patients who made intrauterin surgery.
* Over 40 years of age women.
* Patients with preimplantation genetic diagnosis.
* Anovulatory patient.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — woman who is infertile at reproductive age
Study Population: This study will bw carried out as a prospective randomized clinical trial on regular menstruating patients arriving for transfer of frozen embryo to the center in a single IVF center. Results will collected and recorded daily during the study. With 80% power analysis minimum number of patients 0.05% significance level is 240.
  Study will be designed in 1 year.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
birth | bigger than 24 weeks pregnancy
  live birth

SECONDARY OUTCOMES:
pregnancy rate | 10th day after embryo transfer
  hcg blood test
clinical pregnancy rate | 8 weeks
  positive fetal cardiac activity
abortion rate | 8 weeks
  abortion after visualization of fetal cardiac activity

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Aydın, Study Director — acıbadem university atakent hospital; Elif Ganime Aydeniz, Study Chair — acıbadem university atakent hospital; Emine Karabük, Study Chair — acıbadem university atakent hospital; Burak Yücel, Study Chair — Kanuni Sultan SüleymanHospital
Locations (1):
- Acibadem MAA University Atakent Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We did not decide for this but if they need any information we can support all

REFERENCES:
- [Background] Weissman A, Horowitz E, Ravhon A, Steinfeld Z, Mutzafi R, Golan A, Levran D. Spontaneous ovulation versus HCG triggering for timing natural-cycle frozen-thawed embryo transfer: a randomized study. Reprod Biomed Online. 2011 Oct;23(4):484-9. doi: 10.1016/j.rbmo.2011.06.004. Epub 2011 Jun 15. PMID 21840758
- [Background] Groenewoud ER, Cantineau AE, Kollen BJ, Macklon NS, Cohlen BJ. What is the optimal means of preparing the endometrium in frozen-thawed embryo transfer cycles? A systematic review and meta-analysis. Hum Reprod Update. 2013 Sep-Oct;19(5):458-70. doi: 10.1093/humupd/dmt030. Epub 2013 Jul 2. PMID 23820515
- [Result] Kupka MS, Ferraretti AP, de Mouzon J, Erb K, D'Hooghe T, Castilla JA, Calhaz-Jorge C, De Geyter C, Goossens V; European IVF-Monitoring Consortium, for the European Society of Human Reproduction and Embryology. Assisted reproductive technology in Europe, 2010: results generated from European registers by ESHREdagger. Hum Reprod. 2014 Oct 10;29(10):2099-113. doi: 10.1093/humrep/deu175. Epub 2014 Jul 27. PMID 25069504
- [Result] Fatemi HM, Kyrou D, Bourgain C, Van den Abbeel E, Griesinger G, Devroey P. Cryopreserved-thawed human embryo transfer: spontaneous natural cycle is superior to human chorionic gonadotropin-induced natural cycle. Fertil Steril. 2010 Nov;94(6):2054-8. doi: 10.1016/j.fertnstert.2009.11.036. Epub 2010 Jan 25. PMID 20097333